CLINICAL TRIAL: NCT01256723
Title: Multicenter Prospective Registry of PCI With a New Generation Everolimus- Eluting Stent for Unprotected Left Main Coronary Artery Disease
Brief Title: Japan Unprotected Left Main Coronary Artery Disease Percutaneous Coronary Intervention (PCI) Strategy On New Generation Stents
Acronym: J-LESSON
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Responsible Party: Sponsor
Other Study IDs: J-LESSON2.0
Record Dates: First submitted 2010-11-30; First posted 2010-12-09 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stent (DES); unprotected left main coronary artery (ULMCA)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- J-LESSON Central committee

SUMMARY:
The main purpose of this study is to observe the incidence of major adverse cardiac and cerebrovascular events (MACCE), target vessel failure (TVF), target vessel revascularization (TVR) and stent thrombosis out to 5 years after the procedure in patients who underwent percutaneous coronary intervention (PCI) with everolimus-eluting stents for unprotected left main coronary artery (ULMCA) disease and lesions involving the ULMCA in Japan. The investigators will also establish a method of adjustment to the Japanese version of the SYNTAX score by conducting an assessment using the SYNTAX score recently reported in the US and Europe as well as the EuroSCORE, and by clarifying the differences of PCI procedures and treatment results in Japan with those reported in the US and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 years or older
2. Patients who have signed a written consent
3. Patients who are indicated for percutaneous coronary intervention (PCI)
4. Patients who are considered to be eligible for drug eluting stents
5. Patients who have a de novo lesion to be treated
6. Patients who have ULMCA and lesions involving the ULMCA
7. Patients who can be treated with two of the longest everolimus-eluting stents in one branch
8. Patients who can receive antiplatelet agents for at least 12 months after placement of the drug eluting stent

Exclusion Criteria:

1. Patients who can not fully understand the contents of informed consent of this study
2. Patients who can not provide informed consent because of their mental retardation or language disorder
3. Patients who cannot be followed up for 2 years after the completion of the stent placement
4. Patients who had previously received PCI or coronary artery bypass graft (CABG) for left main coronary artery (LMCA) disease
5. Patients who are scheduled to undergo cardiac surgery
6. Patients who are enrolled in an ongoing registry or clinical trial. Except for a post-marketing study (PMS) that will not influence the result of this study
7. In principal, patients who have participated or are scheduled to participate in another clinical trial related to cardiac blood vessels before completion of the 2-year follow-up period of this study
8. Patients who have a life expectancy of less than 3 years because of a concomitant disease at enrollment
9. Patients who are on home oxygen therapy (HOT)
10. Patients with a serious valvular disease
11. Patients who are on dialysis treatment
12. Patients with severe renal dysfunction (serum creatinine ≥ 2.0 mg/dL)
13. Patients with a low left ventricular ejection fraction of less than 30%
14. Patients with acute myocardial infarction or CK (CPK) levels exceeding twice the institutional upper limit of normal
15. Patients with chronic total occlusions (CTO) in the LMCA
16. Patients who are considered to require a protection device
17. Patients who are confirmed to have an allergy or hypersensitivity to everolimus, acrylic polymer, fluoropolymer or cobalt chrome alloy L-605
18. Patients who have side effects of antiplatelet agents or anticoagulants
19. Nursing women or those of childbearing potential whose pregnancy test conducted within 14 days before the procedure was positive
20. Patients disqualified from participation by the investigator/sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The left coronary artery superintendence part change to a morbid state is possessed, and it is a patient for whom the PCI treatment is necessary.
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac and cerebrovascular events (MACCE) | At 2 years after the procedure
  Incidence of major adverse cardiac and cerebrovascular events (MACCE) at 2 years after the procedure

SECONDARY OUTCOMES:
Assessment of lesions by SYNTAX Score | Baseline procedure
Assessment of lesion by EuroSCORE | Baseline procedure
Assessment of bifurcation lesion by intravascular ultrasound (IVUS) | Baseline procedure
Assessment of bifurcation lesion by intravascular ultrasound (IVUS) | At 10 months post-procedure
Assessment of bifurcation lesion by fractional flow reserve (FFR) | Baseline procedure
Assessment of bifurcation lesion by fractional flow reserve (FFR) | At 10 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, M.D, Study Chair
Locations (1):
- Non-profit organization Associations for Establishment of Evidence in Interventions, Hamamatsuchō, Tokyo, Japan